CLINICAL TRIAL: NCT03337724
Title: A Double-Blind, Placebo-Controlled, Randomized Phase III Study of Ipatasertib in Combination With Paclitaxel as a Treatment for Patients With PIK3CA/AKT1/PTEN-Altered, Locally Advanced or Metastatic, Triple-Negative Breast Cancer or Hormone Receptor-Positive, HER2-Negative Breast Cancer
Brief Title: A Study of Ipatasertib in Combination With Paclitaxel as a Treatment for Participants With PIK3CA/AKT1/PTEN-Altered, Locally Advanced or Metastatic, Triple-Negative Breast Cancer or Hormone Receptor-Positive, HER2-Negative Breast Cancer
Acronym: IPATunity130
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO40016; 2017-001548-36 (EudraCT Number)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ipatasertib + Paclitaxel (Experimental)
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Placebo + Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib, 400 milligrams (mg), administered orally once a day (QD) on Days 1-21 of each 28-day cycle until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
  Arms: Ipatasertib + Paclitaxel
Drug: Paclitaxel — Paclitaxel, 80 mg/square meter (m^2), administered intravenously (IV) on Days 1, 8, and 15 of each 28-day cycle until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
Drug: Placebo — Matching placebo, administered orally QD on Days 1-21 of each 28-day cycle until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
  Arms: Placebo + Paclitaxel

SUMMARY:
This study will evaluate the efficacy of ipatasertib + paclitaxel versus placebo + paclitaxel in participants with histologically confirmed, locally advanced or metastatic triple-negative breast cancer (TNBC) and in participants with locally advanced or metastatic hormone receptor positive (HR+)/ human epidermal growth factor receptor 2 negative (HER2-) breast adenocarcinoma who are not suitable for endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women or men aged =>18 years with histologically documented triple-negative breast cancer (TNBC) or HR+/HER2- adenocarcinoma of the breast that is locally advanced or metastatic and is not amenable to resection with curative intent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate hematologic and organ function within 14 days prior to treatment initiation
* Histologically documented TNBC or HR+/HER2- adenocarcinoma of the breast that is locally advanced or metastatic and is not amenable to resection with curative intent
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eligible for taxane monotherapy, as per local investigator assessment (e.g., absence of rapid clinical progression, life-threatening visceral metastases, or the need for rapid symptom and/or disease control which may require combination chemotherapy)
* HR+/HER2- breast cancer that is not considered appropriate for endocrine-based therapy and meets one of the following: patient has recurrent disease <=5 years of being on adjuvant endocrine therapy or if patient with de novo metastatic disease have progressed within 6 months of being on first line endocrine therapy.
* Consent to submit a formalin-fixed, paraffin-embedded tumor (FFPE) tissue block or freshly cut unstained, serial tumor slides from the most recently collected tumor tissue for central molecular analysis
* Confirmation of biomarker eligibility using an appropriately validated molecular assay at a diagnostic laboratory, Clinically Laboratory Improvement Amendments (CLIA) or equivalently accredited i.e., valid results from either central testing or local testing of tumor tissue or blood demonstrating PIK3CA/AKT1/PTEN-altered status
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods and agreement to refrain from donating sperm

Exclusion Criteria:

* Treatment with approved or investigational cancer therapy within 14 days prior to treatment initiation
* Any previous chemotherapy for inoperable locally advanced or metastatic TNBC or HR+/HER2- adenocarcinoma of the breast (patients receiving neo/adjuvant chemotherapy eligible provided they have at least a 12 month disease-free interval)
* History of or known presence of brain or spinal cord metastases
* Malignancies other than breast cancer within 5 years prior to treatment initiation (except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer)
* Prior treatment with an Akt inhibitor (prior PI3K or mTOR inhibitors are allowed)
* History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills
* Active infection requiring systemic anti-microbial treatment (including antibiotics, anti-fungals, and anti-viral agents)
* Known human immunodeficiency virus (HIV) infection
* Known clinically significant history of liver disease consistent with Child-Pugh Class B or C, including active viral or other hepatitis, current drug or alcohol abuse, or cirrhosis
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of treatment (or anticipated need during study)
* Pregnant or breastfeeding, or intending to become pregnant during the study
* Clinically significant cardiac dysfunction (including NYHA Class II/III/IV heart failure, left ventricular ejection fraction [LVEF] <50%, active ventricular arrhythmia requiring medication, history of myocardial infarction within 6 months of treatment initiation, clinically significant electrocardiogram [ECG] abnormalities).
* Need for chronic corticosteroid therapy of >=10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressants for a chronic disease
* Unresolved, clinically significant toxicity from prior therapy, except for alopecia and Grade 1 peripheral neuropathy
* Uncontrolled clinical symptoms including pleural effusion, pericardial effusion, or ascites, tumor-related pain, hypercalcemia (or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy)
* History of Type I or Type II diabetes mellitus requiring insulin
* Grade >=2 uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia
* History of or active inflammatory bowel disease or active bowel inflammation
* Clinically significant lung disease (including pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, active infection/ history of opportunistic infections)
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of treatment
* Grade >=2 peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (176):
- United States (28):
  - UCSD Moores Cancer Center, La Jolla, California
  - USC Norris Cancer Center, Los Angeles, California
  - USC Norris Cancer Center; USC Oncology Hematology Newport Beach, Newport Beach, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Kaiser Permanente - Roseville, Roseville, California
  - UC Davis; Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente - San Francisco (2238 Geary), San Francisco, California
  - UCSF Comprehensive Cancer Ctr, San Francisco, California
  - K. Permanente - San Jose, San Jose, California
  - Kaiser Permanente - San Leandro, San Leandro, California
  - K. Permanente - Santa Clara, Santa Clara, California
  - Kaiser Permanente - South San Francisco, South San Francisco, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - K. Permanente - Walnut Creek, Walnut Creek, California
  - Memorial Regional Hospital, Hollywood, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - University of Maryland, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - Memorial Sloan Kettering, New York, New York
  - West Clinic, Germantown, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - UT Southwestern Medical Center; Simmons Comprehensive Cancer Center, Simmons Pharmacy, Dallas, Texas
  - Oncology Consultants PA, Houston, Texas
- Argentina (2):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Hosp Provincial D. Centenarios; Oncology Dept, Rosario
- Australia (6):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Westmead Hospital; Medical Oncology, Wentworthville, New South Wales
  - Mater Hospital; Cancer Services, South Brisbane, Queensland
  - Cabrini Medical Centre; Oncology, Malvern, Victoria
  - Fiona Stanley Hospital; FSH Cancer Centre Clinical Trials Unit, Bull Creek, Western Australia
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Notre Dame, Charleroi
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (8):
  - Santa Casa de Misericordia de Salvador, Salvador, Estado de Bahia
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital do Câncer de Londrina, Londrina, Paraná
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
- Canada (2):
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - Jewish General Hospital, Montreal, Quebec
- Sociedad de Investigaciones Medicas Ltda (SIM), Temuco, Chile
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- Czechia (2):
  - Masaryk?v onkologický ústav; Klinika komplexní onkologické pé?e, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
- France (7):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - ICM; Medecine B3, Montpellier
  - Centre Catherine De Sienne, Nantes
  - APHP - Hospital Saint Louis, Paris
  - Institut Jean Godinot; Oncologie Medicale, Reims
- Germany (10):
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Praxis Dr.med. Katja Ziegler-Löhr, Cologne
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf; Frauenklinik, Hamburg
  - Universitätsklinikum des Saarlandes; Klinik f. Frauenheilkunden und Geburtshilfe, Homburg/Saar
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - Mühlenkreiskliniken; Johannes Wesling Klinikum Minden; Klinik für Frauenheilkunde und Geburtshilfe, Minden
  - Oncologianova GmbH - Gesellschaft für Innovationen in der Onkologie, Recklinghausen
  - Universitätsfrauen- und Poliklinik am Klinikum Suedstadt, Rostock
  - Universitätsklinikum Würzburg; Frauenklinik, Würzburg
- Greece (3):
  - Anticancer Hospital Ag Savas; 1St Dept of Internal Medicine, Athens
  - Agioi Anargyroi; 3Rd Dept. of Medical Oncology, Athens
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
- Hungary (5):
  - Orszagos Onkologial Intezet; Onkologiai Osztaly X, Budapest
  - Borsod-Abauj-Zemplen Megyei Korhaz Es Egyetemi Oktato Korhaz; Onkologiai Osztaly, Miskolc
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
  - Hetenyi Geza County Hospital; Onkologiai Kozpont, Szolnok
  - Zala County Hospital ICU, Zalaegerszeg
- India (2):
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Inst.&Research Center; Medical Oncology, New Delhi, National Capital Territory of Delhi
- Italy (5):
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE;U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Ospedale Santa Maria Annunziata; Oncologia, Bagno a Ripoli, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto
- Japan (19):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Kyushu Cancer Center;Breast Oncology, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hyogo Medical University Hospital, Hyōgo
  - St. Marianna University Hospital, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kumamoto Shinto General Hospital, Kumamoto
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Kinki University Hospital, Faculty of Medicine; Surgery, Osaka
  - Saitama Cancer Center, Breast Oncology, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Showa University Hospital; Breast Surgery, Tokyo
- Mexico (4):
  - Centro Medico Dalinde, Mexico City, Mexico CITY (federal District)
  - Centro Médico Zambrano Hellion, Monterrey, Nuevo León
  - Merida | Investigacion Clinica, Mérida, Yucatán
  - CENEIT Oncologicos; DENTRO DE CONDOMINIO SAN FRANCISCO, Mexico City
- North Macedonia (3):
  - Clinical Hospital; Oncology Department, Bitola
  - PHI University Clinic of Radiotherapy and Oncology; Breast malignancy, Skopje
  - PHI University Clinic of Radiotherapy and Oncology; Malignant diseases of thorax, Skopje
- Peru (8):
  - Centro Medico Monte Carmelo, Arequipa
  - Hospital Daniel Alcides Carrion, Callao
  - Clínica San Gabriel; Unidad de Investigación Oncológica de la Clínica San Gabriel, Lima
  - Hospital Nacional Cayetano Heredia; Ocología; Servicio de Hematología Oncología Médica, Lima
  - Oncosalud Sac; Oncología, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clinica Ricardo Palma, San Isidro
  - Instituto Regional de Enfermedades Neoplasicas - IREN Norte, Trujillo
- Poland (3):
  - Instyt. Centrum Zdrowia Matki Polki; Klinika Chirurgii Onk. Chorób Piersi z Podod. Onko Klinicznej, ?ód?
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice; III Klin. Radioter. i Chemioter., Gliwice
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie; Klinika Nowotworow Piersi i Chirurgii Rekonstr, Warsaw
- Russia (9):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Federal State Institution, Moscow Research Oncology Institute n.a. P.A. Hertzen; Oncourology, Moscow, Moscow Oblast
  - Blokhin Cancer Research Center; Combined Treatment, Moskva, Moscow Oblast
  - FSI Rostov research oncological institute of MoH and SD of RF; PAD, Rostov-on-Don, Rostov Oblast
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan', Tatarstan Republic
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - SBIH Kaluga Region Clinical Oncology Dispensary, Kaluga
- Singapore (2):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Medical Oncology Centre of Rosebank; Oncology, Johannesburg, South Africa
- South Korea (7):
  - National Cancer Center, Goyang-si
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (12):
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital de Donostia; Servicio de Oncologia, Guipuzcoa, Guipuzcoa
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic Barcelona; Servicio de oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hospital Clinico Universitario; Oncologia, Valencia
- Taiwan (4):
  - Chi Mei Medical Center Liou Ying Campus, Liuying Township
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - National Taiwan Uni Hospital; General Surgery, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
- Turkey (Türkiye) (6):
  - Ankara Bilkent City Hospital, Ankara
  - Dicle Uni Medical Faculty; Internal Medicine, Diyarbakır
  - Medipol University Medical Faculty; Oncology Department, Istanbul
  - Prof. Dr. Cemil Tascioglu City Hospital; Med Onc, Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital; Oncology, Izmir
  - Sakarya University Medical School; Medical Oncology, Sakarya
- Ukraine (4):
  - Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk
  - Kyiv City Clinical Oncological Center, Day Hospital Department for Oncological patients, Kiev
  - National Cancer Institute MOH of Ukraine, Kiev
  - Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv
- United Kingdom (7):
  - Velindre Cancer Centre, Cardiff
  - University Hospital coventry; Oncology Department, Coventry
  - The Beatson West of Scotland Cancer Centre; Cancer Clinical Trials Unit, Glasgow
  - Royal Marsden Hospital - London, London
  - Derriford Hospital, Plymouth
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Turner N, Dent RA, O'Shaughnessy J, Kim SB, Isakoff SJ, Barrios C, Saji S, Bondarenko I, Nowecki Z, Lian Q, Reilly SJ, Hinton H, Wongchenko MJ, Kovic B, Mani A, Oliveira M. Ipatasertib plus paclitaxel for PIK3CA/AKT1/PTEN-altered hormone receptor-positive HER2-negative advanced breast cancer: primary results from cohort B of the IPATunity130 randomized phase 3 trial. Breast Cancer Res Treat. 2022 Feb;191(3):565-576. doi: 10.1007/s10549-021-06450-x. Epub 2021 Dec 3. PMID 34860318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with protocol specified triple-negative breast cancer (TNBC) or HR+/HER- took part in the study in the following countries: Argentina, Australia, Belgium, Brazil, Canada, Chile, Costa Rica, Czech Republic, France, Greece, Germany, Hungary, Italy, India, Japan, Macedonia, Mexico, Poland, Peru, Republic of Korea, Russian Federation, Slovenia, Spain, Singapore, South Africa, Taiwan, Turkey, Ukraine, United Kingdom, and United States from 6 January 2018 to 4 January 2023.
Pre-assignment Details: Participants with TNBC or hormone receptor positive(HR+)/human epidermal growth factor receptor 2 negative(HER2-) breast adenocarcinoma with phosphatidylinositol-4,5-bisphosphate3-kinase,catalytic subunit, alpha(PIK3CA)/serine-threonine kinase(AKT1)/phosphatase & tensin homolog (PTEN)-altered tumor were randomized to ipatasertib 400 mg+paclitaxel or placebo+paclitaxel (Cohorts A,B) & those with TNBC without PIK3CA/ AKT1/PTEN-altered tumor received ipatasertib+atezolizumab+paclitaxel (Cohort C).
Groups:
- Cohort A: Placebo + Paclitaxel: Participants with histologically confirmed locally advanced unresectable or metastatic TNBC with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 milligram per square meter (mg/m^2), intravenously (IV), on Days 1, 8, and 15 of each 28-day cycle and placebo, orally once a day (QD), on Days 1 to 21 of each 28-day cycle up to 58.9 months.
- Cohort A: Ipatasertib + Paclitaxel: Participants with histologically confirmed locally advanced unresectable or metastatic TNBC with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, at a dose of 400 mg, administered orally QD, on Days 1 to 21 of each 28-day cycle up to 58.9 months.
- Cohort B: Placebo + Paclitaxel: Participants with histologically confirmed HR+ /HER2- adenocarcinoma of the breast with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and placebo, orally QD, on Days 1 to 21 of each 28-day cycle up to 59.9 months.
- Cohort B: Ipatasertib + Paclitaxel: Participants with histologically confirmed HR+/HER2- adenocarcinoma of the breast with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, at a dose of 400 mg, administered orally QD, on Days 1 to 21 of each 28-day cycle up to 59.9 months.
- Cohort C: Ipatasertib + Atezolizumab + Paclitaxel: Participants with histologically confirmed locally advanced unresectable or metastatic TNBC without PIK3CA/AKT1/PTEN-altered tumors and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle, ipatasertib at a dose of 400 mg, administered orally QD, on Days 1 to 21 of each 28-day cycle, and atezolizumab 840 mg, IV, on Days 1 and 15 of each 28-day cycle up to 45.5 months.
Period: Overall Study
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Started | 87 | 168 | 76 | 146 | 102
Safety Evaluable Population (Safety Evaluable Population included all participants who received any amount of study treatment. Participants who were randomized (Cohorts A and B) or enrolled (Cohort C) into the study but who did not receive any study drug were not included in the Safety Evaluable Population.) | 87 | 166 | 75 | 145 | 102
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 87 | 168 | 76 | 146 | 102
Not completed — Reason not Specified | 12 | 21 | 9 | 9 | 29
Not completed — Withdrawal by Subject | 13 | 15 | 4 | 15 | 6
Not completed — Protocol Deviation | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0
Not completed — Death | 40 | 89 | 43 | 76 | 50
Not completed — Lost to Follow-up | 5 | 5 | 4 | 7 | 4
Not completed — Physician Decision | 16 | 34 | 14 | 34 | 13
Not completed — Progressive Disease | 0 | 2 | 1 | 2 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) Population included all randomized participants in Cohorts A and B regardless of whether the participants received the assigned treatment. For Cohort C, the ITT population consisted of all enrolled participants in Cohort C.
Groups:
- Cohort A: Placebo + Paclitaxel: Participants with histologically confirmed locally advanced unresectable or metastatic TNBC with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and placebo, orally QD, on Days 1 to 21 of each 28-day cycle up to 58.9 months.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel | Total
Number analyzed (Participants) | 87 | 168 | 76 | 146 | 102 | 579
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (12.6) | 54.6 (12.8) | 54.5 (11.3) | 57.2 (11.1) | 54.6 (11.7) | 55.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 167 | 76 | 144 | 102 | 576
  Male | 0 | 1 | 0 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 59 | 13 | 29 | 36 | 166
  Not Hispanic or Latino | 57 | 101 | 62 | 115 | 58 | 393
  Unknown or Not Reported | 1 | 8 | 1 | 2 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 15 | 3 | 4 | 5 | 40
  Asian | 17 | 37 | 22 | 38 | 12 | 126
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 5 | 3 | 2 | 9 | 20
  White | 51 | 99 | 45 | 93 | 55 | 343
  More than one race | 0 | 4 | 2 | 0 | 5 | 11
  Unknown or Not Reported | 5 | 8 | 1 | 9 | 15 | 38

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression, as determined locally by the investigator through the use of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1), or death from any cause, whichever occurred first, assessed up to 27 months for this outcome measure. Progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions was also considered progression.
Time Frame: From randomization up to 27 months
Population: ITT Population included all randomized participants in Cohorts A regardless of whether the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 87 | 168
months | 6.1 [5.5 to 9.0] | 7.4 [5.6 to 8.5]
Statistical Analysis 1: Comparison: Cohort A: Placebo + Paclitaxel vs Cohort A: Ipatasertib + Paclitaxel; Test type: Superiority; p = 0.9237, Log Rank; Stratified Hazard Ratio = 1.02, 95% CI 2-sided [0.71 to 1.45] — Stratification variables were: prior adjuvant/neoadjuvant chemotherapy (yes vs. no), region, tumor PIK3CA/AKT1/PTEN alteration status (PIK3CA/AKT1-activating mutations vs. PTEN alterations with no PIK3CA/AKT1-activating mutations)

2. Primary Outcome: Cohort B: PFS
Description: PFS was defined as the time from randomization to the first occurrence of disease progression, as determined locally by the investigator through the use of RECIST v.1.1, or death from any cause, whichever occurred first, assessed up to 24.4 months for this outcome measure. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Abbreviation used in statistical analysis: PI3K=phosphoinositide 3-kinase and mTOR=mammalian target of rapamycin inhibitor.
Time Frame: From randomization up to 24.4 months
Population: ITT Population included all randomized participants in Cohort B regardless of whether the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 76 | 146
months | 9.3 [7.2 to 12.2] | 9.3 [8.0 to 11.0]
Statistical Analysis 1: Comparison: Cohort B: Placebo + Paclitaxel vs Cohort B: Ipatasertib + Paclitaxel; Test type: Superiority; p = 0.9965, Log Rank; Stratified Hazard Ratio = 1.00, 95% CI 2-sided [0.71 to 1.40] — Stratification variables were: prior adjuvant/neoadjuvant chemotherapy (yes vs. no), region, prior therapy with a PI3K or mTOR inhibitor (yes vs. no)

3. Primary Outcome: Cohort C: PFS
Description: PFS for Cohort C was defined as the time from enrollment to the first occurrence of disease progression, as determined locally by the investigator through the use of RECIST v.1.1, or death from any cause, whichever occurred first, assessed up to 31 months for this outcome measure. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From enrollment up to 31 months
Population: ITT population included of all enrolled participants in Cohort C.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 102
months | 7.1 [5.5 to 9.1]

4. Secondary Outcome: Cohort A and B: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants with partial response (PR) or complete response (CR) on 2 consecutive occasions ≥4 weeks apart as determined by the investigator using RECIST v.1.1, assessed up to 27 months for Cohort A and up to 24.4 months for Cohort B, for this outcome measure. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Percentages are rounded off to the nearest decimal point.
Time Frame: From randomization up to 27 months for Cohort A and up to 24.4 months for Cohort B
Population: ITT Population included all randomized participants in Cohorts A and B regardless of whether the participants received the assigned treatment. Overall number analyzed is the number of participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 86 | 167 | 75 | 144
percentage of participants | 34.9 [24.92 to 45.92] | 38.9 [31.49 to 46.76] | 46.7 [35.05 to 58.55] | 46.5 [38.18 to 55.02]

5. Secondary Outcome: Cohort C: ORR
Description: ORR was defined as percentage of participants with PR or CR on 2 consecutive occasions ≥4 weeks apart as determined by the investigator using RECIST v.1.1, assessed up to 31 months for this outcome measure. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. Percentages are rounded off to the nearest decimal point.
Time Frame: From enrollment up to 31 months
Population: ITT population consisted of all enrolled participants in Cohort C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 102
percentage of participants | 52.9 [42.80 to 62.90]

6. Secondary Outcome: Cohort A and B: Duration of Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented OR (CR or PR) to PD, as determined locally by the investigator through the use of RECIST v1.1, or death from any cause, whichever occurred first assessed up to 27 months for Cohort A and up to 24.4 months for Cohort B, for this outcome measure. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From randomization up to 27 months for Cohort A and up to 24.4 months for Cohort B
Population: ITT Population included all randomized participants in Cohorts A and B regardless of whether the participants received the assigned treatment. Overall number analyzed is the number of participants with objective response i.e., responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 30 | 65 | 35 | 67
months | 16.6 [4.9 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with event. | 9.4 [7.3 to 11.1] | 9.2 [6.8 to 12.5] | 9.2 [7.2 to 11.3]

7. Secondary Outcome: Cohort C: DOR
Description: DOR was defined as the time from the first occurrence of a documented OR (CR or PR) to PD, as determined locally by the investigator through the use of RECIST v1.1, or death from any cause, whichever occurred first, assessed up to 31 months for this outcome measure. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: From enrollment up to 31 months
Population: ITT population consisted of all enrolled participants in Cohort C. Overall number analyzed is the number of participants with objective response i.e., responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 54
months | 8.7 [5.7 to 12.7]

8. Secondary Outcome: Cohort A and B: Clinical Benefit Rate (CBR)
Description: CBR was defined as percentage of participants with an objective response (CR or PR), or stable disease (SD) for at least 24 weeks, as determined by the investigator through the use of RECIST v.1.1. assessed up to From randomization up to 27 months for Cohort A and up to 24.4 months for Cohort B for this outcome measure. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Percentages are rounded off to the nearest decimal point.
Time Frame: From randomization up to 27 months for Cohort A and up to 24.4 months for Cohort B
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 86 | 167 | 75 | 144
percentage of participants | 45.3 [34.58 to 56.45] | 46.7 [38.96 to 54.57] | 65.3 [53.46 to 75.96] | 68.8 [60.50 to 76.21]

9. Secondary Outcome: Cohort C: CBR
Description: CBR was defined as percentage of participants with an objective response (CR or PR), or SD for at least 24 weeks, as determined by the investigator through the use of RECIST v.1.1 assessed up to 31 months for this outcome measure. CR was defined as the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Percentages are rounded off to the nearest decimal point.
Time Frame: From enrollment up to 31 months
Population: ITT population consisted of all enrolled participants in Cohort C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 102
percentage of participants | 54.9 [44.74 to 64.78]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: From randomization/ enrollment (Cohort C) up to death from any cause, up to 45 months for Cohort A, up to 46 months for Cohort B and up to 31 months for Cohort C
Population: ITT Population included all randomized participants in Cohorts A and B regardless of whether the participants received the assigned treatment. For Cohort C, the ITT population consisted of all enrolled participants in Cohort C.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 87 | 168 | 76 | 146 | 102
months | 24.9 [16.9 to 40.4] | 24.2 [19.2 to 29.4] | 28.4 [20.6 to 37.3] | 29.0 [22.4 to 34.8] | 22.8 [17.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Cohort A: Placebo + Paclitaxel vs Cohort A: Ipatasertib + Paclitaxel; Test type: Superiority; Stratified Hazard Ratio = 1.08, 95% CI 2-sided [0.73 to 1.58] — Stratification was done prior adjuvant/neoadjuvant chemotherapy (yes vs. no), region, tumor PIK3CA/AKT1/PTEN alteration status (PIK3CA/AKT1-activating mutations vs. PTEN alterations with no PIK3CA/AKT1-activating mutations)
Statistical Analysis 2: Comparison: Cohort B: Placebo + Paclitaxel vs Cohort B: Ipatasertib + Paclitaxel; Test type: Superiority; Stratified Hazard Ratio = 0.94, 95% CI 2-sided [0.65 to 1.37] — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: Cohort A and B: Change From Baseline in Global Health Status (GHS)/Health-Related Quality of Life (HRQoL) Score Measured by GHS/HRQoL Scale (Questions 29 and 30) of the EORTC QLQ-C30
Description: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) is a cancer-specific instrument with 30 questions covering symptoms, functioning, and health-related quality of life (HRQoL). The participant's assessment of overall HRQoL is assessed by using the last 2 questions (29 and 30) of the instrument, with each of these items based on a 7-point scale (1=very poor to 7=excellent), which are then combined into the GHS/QoL multi-item scale. The scores obtained for each question were averaged into a raw score for the scale, and this raw score for the scale was then subsequently linearly transformed to a scale score of 0 to 100, with a high score indicating better GHS/QoL. Negative change from Baseline values in the GHS/QoL change from baseline analysis indicated deterioration in HRQoL and positive values indicated improvement.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24 (cycle length=28 days)
Population: Patient-reported outcome (PRO)-evaluable Population included all randomized (Cohorts A and B) participants who had a baseline and at least 1 postbaseline PRO assessment.Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 79 | 160 | 73 | 146
score on scale
  Day 1 Cycle 2: number analyzed (Participants) | 79 | 160 | 73 | 127
  Day 1 Cycle 2 | 0.95 (20.59) | -0.26 (24.58) | 4.79 (15.83) | -3.61 (21.45)
  Day 1 Cycle 3: number analyzed (Participants) | 72 | 143 | 70 | 121
  Day 1 Cycle 3 | -0.93 (20.53) | 0.35 (21.73) | 1.19 (19.62) | -2.13 (17.99)
  Day 1 Cycle 4: number analyzed (Participants) | 62 | 124 | 63 | 113
  Day 1 Cycle 4 | -4.44 (19.42) | -2.42 (21.95) | -0.79 (21.10) | -1.99 (20.75)
  Day 1 Cycle 5: number analyzed (Participants) | 56 | 93 | 56 | 108
  Day 1 Cycle 5 | -2.08 (16.46) | -2.87 (18.61) | -1.19 (20.00) | -3.01 (18.70)
  Day 1 Cycle 6: number analyzed (Participants) | 48 | 77 | 53 | 101
  Day 1 Cycle 6 | -6.94 (15.97) | -2.06 (21.04) | 1.42 (19.18) | -3.88 (20.67)
  Day 1 Cycle 7: number analyzed (Participants) | 35 | 61 | 49 | 94
  Day 1 Cycle 7 | -5.48 (12.45) | -3.28 (20.93) | 0.34 (20.34) | -4.17 (19.47)
  Day 1 Cycle 8: number analyzed (Participants) | 29 | 51 | 48 | 89
  Day 1 Cycle 8 | -6.90 (13.56) | 0.33 (22.11) | 0.35 (16.84) | -5.99 (18.55)
  Day 1 Cycle 9: number analyzed (Participants) | 22 | 43 | 38 | 78
  Day 1 Cycle 9 | 0.00 (10.29) | -3.49 (25.28) | 1.10 (18.80) | -7.37 (20.05)
  Day 1 Cycle 10: number analyzed (Participants) | 21 | 35 | 39 | 70
  Day 1 Cycle 10 | -2.38 (9.91) | -4.52 (21.61) | 1.28 (19.64) | -6.43 (18.83)
  Day 1 Cycle 11: number analyzed (Participants) | 17 | 28 | 35 | 65
  Day 1 Cycle 11 | -3.43 (15.88) | -4.46 (21.09) | 2.38 (22.83) | -5.13 (19.30)
  Day 1 Cycle 12: number analyzed (Participants) | 11 | 23 | 31 | 58
  Day 1 Cycle 12 | 0.76 (11.46) | -8.33 (19.94) | 0.00 (22.46) | -4.02 (16.32)
  Day 1 Cycle 13: number analyzed (Participants) | 8 | 19 | 24 | 43
  Day 1 Cycle 13 | -5.21 (10.85) | -8.33 (23.57) | -2.43 (21.63) | -4.65 (18.57)
  Day 1 Cycle 14: number analyzed (Participants) | 7 | 14 | 22 | 38
  Day 1 Cycle 14 | -2.38 (10.45) | -3.57 (19.26) | -0.76 (21.81) | -3.29 (15.68)
  Day 1 Cycle 15: number analyzed (Participants) | 6 | 13 | 15 | 27
  Day 1 Cycle 15 | -9.72 (11.08) | -5.77 (12.90) | -2.22 (18.49) | -0.62 (20.14)
  Day 1 Cycle 16: number analyzed (Participants) | 5 | 11 | 14 | 25
  Day 1 Cycle 16 | -6.67 (13.69) | -8.33 (14.91) | -4.17 (19.27) | -2.33 (16.05)
  Day 1 Cycle 17: number analyzed (Participants) | 4 | 11 | 12 | 21
  Day 1 Cycle 17 | -8.33 (9.62) | -6.82 (13.34) | -7.64 (15.27) | -5.95 (13.73)
  Day 1 Cycle 18: number analyzed (Participants) | 4 | 7 | 9 | 14
  Day 1 Cycle 18 | -8.33 (9.62) | -15.48 (16.96) | -9.26 (19.74) | -6.55 (16.07)
  Day 1 Cycle 19: number analyzed (Participants) | 4 | 5 | 5 | 12
  Day 1 Cycle 19 | -4.17 (8.33) | -20.00 (7.45) | -11.67 (16.24) | -7.64 (23.96)
  Day 1 Cycle 20: number analyzed (Participants) | 2 | 3 | 4 | 10
  Day 1 Cycle 20 | -8.33 (11.79) | -5.56 (9.62) | -16.67 (11.79) | -10.00 (12.30)
  Day 1 Cycle 21: number analyzed (Participants) | 1 | 2 | 3 | 7
  Day 1 Cycle 21 | -16.67 (NA) — The standard deviation was not estimable for a single participant. | -16.67 (0.00) | -13.89 (20.97) | -10.71 (13.36)
  Day 1 Cycle 22: number analyzed (Participants) | 1 | 1 | 3 | 7
  Day 1 Cycle 22 | -16.67 (NA) — The standard deviation was not estimable for a single participant. | -16.67 (NA) — The standard deviation was not estimable for a single participant. | -11.11 (9.62) | -14.29 (15.00)
  Day 1 Cycle 23: number analyzed (Participants) | 1 | 1 | 3 | 5
  Day 1 Cycle 23 | -16.67 (NA) — The standard deviation was not estimable for a single participant. | -25.00 (NA) — The standard deviation was not estimable for a single participant. | -16.67 (16.67) | -15.00 (18.07)
  Day 1 Cycle 24: number analyzed (Participants) | 1 | 1 | 2 | 2
  Day 1 Cycle 24 | -16.67 (NA) — The standard deviation was not estimable for a single participant. | -41.67 (NA) — The standard deviation was not estimable for a single participant. | -16.67 (0.00) | -16.67 (11.79)

12. Secondary Outcome: Cohort C: Change From Baseline in GHS/HRQoL Score Measured by GHS/HRQoL Scale (Questions 29 and 30) of the EORTC QLQ-C30
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions covering symptoms, functioning, and health-related quality of life (HRQoL). The participant's assessment of overall HRQoL is assessed by using the last 2 questions (29 and 30) of the instrument, with each of these items based on a 7-point scale (1=very poor to 7=excellent), which are then combined into the GHS/QoL multi-item scale. The scores obtained for each question were averaged into a raw score for the scale, and this raw score for the scale was then subsequently linearly transformed to a scale score of 0 to 100, with a high score indicating better GHS/QoL. Negative change from Baseline values in the GHS/QoL change from baseline analysis indicated deterioration in HRQoL and positive values indicated improvement.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 38, 39, 40, 41, 42, 43, and 44 (cycle length=28 days)
Population: PRO-evaluable Population for Cohort C included all enrolled participants who had a baseline and at least 1 postbaseline PRO assessment.Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 100
score on scale
  Day 1 Cycle 2 | -0.42 (18.02)
  Day 1 Cycle 3: number analyzed (Participants) | 92
  Day 1 Cycle 3 | 0.18 (18.32)
  Day 1 Cycle 4: number analyzed (Participants) | 84
  Day 1 Cycle 4 | -4.37 (22.83)
  Day 1 Cycle 5: number analyzed (Participants) | 65
  Day 1 Cycle 5 | -6.41 (20.19)
  Day 1 Cycle 6: number analyzed (Participants) | 61
  Day 1 Cycle 6 | -7.10 (21.24)
  Day 1 Cycle 7: number analyzed (Participants) | 54
  Day 1 Cycle 7 | -5.09 (18.20)
  Day 1 Cycle 8: number analyzed (Participants) | 50
  Day 1 Cycle 8 | -4.83 (21.24)
  Day 1 Cycle 9: number analyzed (Participants) | 37
  Day 1 Cycle 9 | -7.66 (23.68)
  Day 1 Cycle 10: number analyzed (Participants) | 33
  Day 1 Cycle 10 | -7.07 (18.76)
  Day 1 Cycle 11: number analyzed (Participants) | 25
  Day 1 Cycle 11 | -6.00 (19.02)
  Day 1 Cycle 12: number analyzed (Participants) | 23
  Day 1 Cycle 12 | -2.90 (18.57)
  Day 1 Cycle 13: number analyzed (Participants) | 23
  Day 1 Cycle 13 | -1.45 (19.08)
  Day 1 Cycle 14: number analyzed (Participants) | 19
  Day 1 Cycle 14 | -7.89 (21.24)
  Day 1 Cycle 15: number analyzed (Participants) | 18
  Day 1 Cycle 15 | -5.09 (26.37)
  Day 1 Cycle 16: number analyzed (Participants) | 16
  Day 1 Cycle 16 | -11.98 (27.55)
  Day 1 Cycle 17: number analyzed (Participants) | 13
  Day 1 Cycle 17 | -10.90 (32.16)
  Day 1 Cycle 18: number analyzed (Participants) | 13
  Day 1 Cycle 18 | -3.85 (20.30)
  Day 1 Cycle 19: number analyzed (Participants) | 13
  Day 1 Cycle 19 | -3.21 (25.35)
  Day 1 Cycle 20: number analyzed (Participants) | 13
  Day 1 Cycle 20 | -3.21 (24.89)
  Day 1 Cycle 21: number analyzed (Participants) | 13
  Day 1 Cycle 21 | -2.56 (24.86)
  Day 1 Cycle 22: number analyzed (Participants) | 13
  Day 1 Cycle 22 | -12.18 (32.92)
  Day 1 Cycle 23: number analyzed (Participants) | 11
  Day 1 Cycle 23 | 3.03 (24.23)
  Day 1 Cycle 24: number analyzed (Participants) | 11
  Day 1 Cycle 24 | 3.79 (24.54)
  Day 1 Cycle 25: number analyzed (Participants) | 9
  Day 1 Cycle 25 | -4.63 (21.29)
  Day 1 Cycle 26: number analyzed (Participants) | 10
  Day 1 Cycle 26 | -0.83 (19.82)
  Day 1 Cycle 27: number analyzed (Participants) | 8
  Day 1 Cycle 27 | 2.08 (26.63)
  Day 1 Cycle 28: number analyzed (Participants) | 6
  Day 1 Cycle 28 | 1.39 (23.81)
  Day 1 Cycle 29: number analyzed (Participants) | 7
  Day 1 Cycle 29 | -1.19 (28.64)
  Day 1 Cycle 30: number analyzed (Participants) | 5
  Day 1 Cycle 30 | 3.33 (24.01)
  Day 1 Cycle 31: number analyzed (Participants) | 3
  Day 1 Cycle 31 | 22.22 (12.73)
  Day 1 Cycle 32: number analyzed (Participants) | 4
  Day 1 Cycle 32 | 10.42 (23.94)
  Day 1 Cycle 33: number analyzed (Participants) | 3
  Day 1 Cycle 33 | 16.67 (22.05)
  Day 1 Cycle 34: number analyzed (Participants) | 3
  Day 1 Cycle 34 | 16.67 (30.05)
  Day 1 Cycle 35: number analyzed (Participants) | 3
  Day 1 Cycle 35 | 13.89 (17.35)
  Day 1 Cycle 36: number analyzed (Participants) | 2
  Day 1 Cycle 36 | 20.83 (29.46)
  Day 1 Cycle 37: number analyzed (Participants) | 2
  Day 1 Cycle 37 | 16.67 (23.57)
  Day 1 Cycle 38: number analyzed (Participants) | 2
  Day 1 Cycle 38 | 16.67 (23.57)
  Day 1 Cycle 39: number analyzed (Participants) | 2
  Day 1 Cycle 39 | 25.00 (35.36)
  Day 1 Cycle 40: number analyzed (Participants) | 1
  Day 1 Cycle 40 | 33.33 (NA) — The standard deviation was not estimable for a single participant.
  Day 1 Cycle 41: number analyzed (Participants) | 1
  Day 1 Cycle 41 | 50.00 (NA) — The standard deviation was not estimable for a single participant.
  Day 1 Cycle 42: number analyzed (Participants) | 1
  Day 1 Cycle 42 | 41.67 (NA) — The standard deviation was not estimable for a single participant.
  Day 1 Cycle 43: number analyzed (Participants) | 1
  Day 1 Cycle 43 | 41.67 (NA) — The standard deviation was not estimable for a single participant.
  Day 1 Cycle 44: number analyzed (Participants) | 1
  Day 1 Cycle 44 | 50.00 (NA) — The standard deviation was not estimable for a single participant.

13. Secondary Outcome: Cohort B: Time to Deterioration (TTD) in Pain
Description: Time to deterioration in GHS/HRQoL was defined as the time from randomization to first observed ≥ 11-point increase from Baseline in pain scale score (Question 9 and 19) in EORTC QLQ-C30 linearly transformed GHS/HRQoL scale score, assessed up 24.4 months for this outcome measure. TTD was planned to be assessed only in cohort with HR+/HER2 - breast cancer participants (Cohort B). Questions 9 and 19 that assessed pain, used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). The scores were linearly transformed on a scale of 0 to 100, with higher scores indicating increased severity in symptoms.
Time Frame: Baseline up to 24.4 months
Population: ITT Population for Cohort B included as all randomized participants regardless of whether the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 76 | 146
months | NA [NA to NA] — Median and 95% CI were not estimable due to insufficient number of participants with events. | NA [11.1 to NA] — Median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Cohort B: Placebo + Paclitaxel vs Cohort B: Ipatasertib + Paclitaxel; Test type: Superiority; p = 0.2162, Log Rank; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.83 to 2.22] — [estimate comment as in outcome 2, analysis 1]; Stratified Analysis

14. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs were reported based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0.
Time Frame: Up to 58.9 months for Cohort A, up to 59.9 months for Cohort B and up to 45.5 months for Cohort C
Population: Safety Evaluable Population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 87 | 166 | 75 | 145 | 102
Participants | 84 | 162 | 74 | 144 | 102

15. Secondary Outcome: Number of Participants With at Least One Adverse Events of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs were reported based on the NCI CTCAE, Version 4.0. AESI include cases of potential drug-induced liver injury that include an elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law. Suspected transmission of an infectious agent by the study drug, Grade >= 3 fasting hyperglycemia, hepatotoxicity, diarrhea, rash, ALT/AST elevations. Grade >= 2 colitis/enterocolitis.
Time Frame: Up to 58.9 months for Cohort A, up to 59.9 months for Cohort B and up to 45.5 months for Cohort C
Population: Safety Evaluable Population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo + Paclitaxel | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Placebo + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 87 | 166 | 75 | 145 | 102
Participants | 79 | 157 | 73 | 141 | 101

16. Secondary Outcome: Cohorts A and B:Plasma Concentration of Ipatasertib
Time Frame: Days 1 and 15 of Cycle 1: 1 to 3 hours post dose, and on Day 15 of Cycle 3: 2 to 4 hours post dose (cycle length= 28 days)
Population: PK Evaluable Population included all participants who had at least one evaluable plasma sample. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 146 | 132
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 | 176 (232) | 165 (326)
  Cycle 1 Day 15: number analyzed (Participants) | 132 | 119
  Cycle 1 Day 15 | 191 (184) | 211 (216)
  Cycle 3 Day 15: number analyzed (Participants) | 110 | 102
  Cycle 3 Day 15 | 165 (169) | 234 (149)

17. Secondary Outcome: Cohort C: Plasma Concentration of Ipatasertib
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 94
ng/mL
  Cycle 1 Day 1 | 175 (183)
  Cycle 1 Day 15: number analyzed (Participants) | 82
  Cycle 1 Day 15 | 233 (161.6)
  Cycle 3 Day 15: number analyzed (Participants) | 62
  Cycle 3 Day 15 | 207 (197.6)

18. Secondary Outcome: Cohorts A and B: Plasma Concentration of G-037720
Description: G-037720 was a metabolite of ipatasertib.
Time Frame: Days 1 and 15 of Cycle 1: 1 to 3 hours post dose, and on Day 15 of Cycle 3: 2 to 4 hours post dose (cycle length= 28 days )
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: Ipatasertib + Paclitaxel | Cohort B: Ipatasertib + Paclitaxel
Number analyzed (Participants) | 146 | 123
ng/mL
  Cycle 1 Day 1 | 45.6 (777) | 68.2 (405)
  Cycle 1 Day 15: number analyzed (Participants) | 132 | 119
  Cycle 1 Day 15 | 83.9 (183) | 95.1 (211)
  Cycle 3 Day 15: number analyzed (Participants) | 110 | 102
  Cycle 3 Day 15 | 90.8 (180) | 109 (169)

19. Secondary Outcome: Cohort C: Plasma Concentration of G-037720
Description: G-037720 was a metabolite of ipatasertib.
Time Frame: as for outcome 18
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 91
ng/mL
  Cycle 1 Day 1 | 67.3 (222.3)
  Cycle 1 Day 15: number analyzed (Participants) | 82
  Cycle 1 Day 15 | 96.8 (140.7)
  Cycle 3 Day 15: number analyzed (Participants) | 62
  Cycle 3 Day 15 | 96.5 (167.9)

20. Secondary Outcome: Cohort C: 1-year Event-free PFS Rate
Description: PFS was defined as the time from enrollment to the first occurrence of disease progression, as determined locally by the investigator through the use of RECIST v.1.1, or death from any cause, whichever occurred first. Event-free PFS rate was defined as percentage of participants who did not experience any event and survived at 1 year after enrollment. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression. Percentages are rounded off to the nearest decimal point. As prespecified in the protocol, this outcome measure was applicable only to Cohort C.
Time Frame: From enrollment until the occurrence of disease progression or death from any cause, whichever occurred earlier, up to 1 year
Population: ITT Population for Cohort C included all enrolled participants in Cohort C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 102
percentage of participants | 31.17 [21.59 to 40.76]

21. Secondary Outcome: Cohort C: 1-year Event-free OS Rate
Description: OS was defined as the time from enrollment to death from any cause. Event-free OS rate was defined as percentage of participants who did not experience any event and survived at 1 year after enrollment. As prespecified in the protocol, this outcome measure was applicable only to Cohort C. Percentages were rounded off to the nearest decimal.
Time Frame: From enrollment up to death from any cause, up to 1 year
Population: ITT Population for Cohort C included all enrolled participants in Cohort C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 102
percentage of participants | 79.38 [71.31 to 87.44]

22. Secondary Outcome: Cohort C: Serum Concentration of Atezolizumab
Description: As prespecified in the protocol, this outcome measure was applicable only to Cohort C.
Time Frame: Day 1 of Cycle 1: 30 minutes post dose, predose on Day 15 of Cycle 1 and predose on Day 1 of Cycles 2, 3, 4, 8, 12 and 16 (cycle length=28 days)
Population: For Cohort C, PK Evaluable Population included all participants who had at least one evaluable plasma sample in Cohort C. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 101
micrograms per milliliter (µg/mL)
  Day 1 Cycle 1: number analyzed (Participants) | 84
  Day 1 Cycle 1 | 309 (31.7)
  Day 15 Cycle 1: number analyzed (Participants) | 78
  Day 15 Cycle 1 | 91.5 (23.9)
  Day 1 Cycle 2: number analyzed (Participants) | 92
  Day 1 Cycle 2 | 130 (54.1)
  Day 1 Cycle 3: number analyzed (Participants) | 84
  Day 1 Cycle 3 | 200 (41.1)
  Day 1 Cycle 4: number analyzed (Participants) | 80
  Day 1 Cycle 4 | 231 (52.3)
  Day 1 Cycle 8: number analyzed (Participants) | 46
  Day 1 Cycle 8 | 327 (27.6)
  Day 1 Cycle 12: number analyzed (Participants) | 21
  Day 1 Cycle 12 | 371 (30.5)
  Day 1 Cycle 16: number analyzed (Participants) | 12
  Day 1 Cycle 16 | 402 (42.4)

23. Secondary Outcome: Cohort C: Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: The numbers of ADA-positive participants after drug administration were summarized for participants exposed to atezolizumab. As prespecified in the protocol, this outcome measure was applicable only to Cohort C.
Time Frame: Up to 45.5 months
Population: For Cohort C, Safety Evaluable Population included all participants who received any amount of study treatment in cohort C. Overall number analyzed is the number of participants with an ADA assay result from at least one post-baseline sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort C: Ipatasertib + Atezolizumab + Paclitaxel
Number analyzed (Participants) | 101
Participants | 18

ADVERSE EVENTS:
Time Frame: Up to 58.9 months for Cohort A, up to 59.9 months for Cohort B and up to 45.5 months for Cohort C
Description: All-cause Mortality: ITT Population included all randomized participants in Cohorts A and B regardless of whether the participants received the assigned treatment. For Cohort C, the ITT population consisted of all enrolled participants in Cohort C. Serious and Other Adverse Events: Safety Evaluable Population included all participants who received any amount of study treatment.
Groups:
- COHORT A Placebo + Paclitaxel: Participants with histologically confirmed locally advanced unresectable or metastatic TNBC with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and placebo, administered orally QD, on Days 1 to 21 of each 28-day cycle up to 58.9 months.
- COHORT A Ipatasertib + Paclitaxel: Participants with histologically confirmed locally advanced unresectable or metastatic TNBC with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, at a dose of 400 mg, administered orally QD, on Days 1 to 21 of each 28-day cycle up to 58.9 months.
- COHORT B Placebo + Paclitaxel: Participants with histologically confirmed HR+ /HER2- adenocarcinoma of the breast with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and placebo, orally QD, on Days 1 to 21 of each 28-day cycle up to 59.9 months.
- COHORT B Ipatasertib + Paclitaxel: Participants with histologically confirmed HR+/HER2- adenocarcinoma of the breast with PIK3CA/AKT1/PTEN alteration and no prior systemic chemotherapy in the advanced disease setting and who were candidates for taxane monotherapy received paclitaxel chemotherapy, 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, at a dose of 400 mg, administered orally QD, on Days 1 to 21 of each 28-day cycle up to 59.9 months.
- COHORT C Ipatasertib + Atezolizumab + Paclitaxel: Participants with histologically confirmed locally advanced unresectable or metastatic TNBC without PIK3CA/AKT1/PTEN-altered tumors and no prior systemic chemotherapy in the advanced disease setting received paclitaxel chemotherapy 80 mg/m^2, IV, on Days 1, 8, and 15 of each 28-day cycle, ipatasertib at a dose of 400 mg, administered orally QD, on Days 1 to 21 of each 28-day cycle, and atezolizumab 840 mg, IV, on Days 1 and 15 of each 28-day cycle up to 45.5 months.
Arm/Group | COHORT A Placebo + Paclitaxel | COHORT A Ipatasertib + Paclitaxel | COHORT B Placebo + Paclitaxel | COHORT B Ipatasertib + Paclitaxel | COHORT C Ipatasertib + Atezolizumab + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 41/87 | 91/168 | 44/76 | 78/146 | 50/102
Serious Adverse Events (participants affected / at risk) | 20/87 | 34/166 | 11/75 | 30/145 | 29/102
Other Adverse Events (participants affected / at risk) | 82/87 | 161/166 | 72/75 | 141/145 | 101/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT A Placebo + Paclitaxel (N=87) | COHORT A Ipatasertib + Paclitaxel (N=166) | COHORT B Placebo + Paclitaxel (N=75) | COHORT B Ipatasertib + Paclitaxel (N=145) | COHORT C Ipatasertib + Atezolizumab + Paclitaxel (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (8) | 1 (1) | 4 (5) | 4 (4)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emphysematous cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT A Placebo + Paclitaxel (N=87) | COHORT A Ipatasertib + Paclitaxel (N=166) | COHORT B Placebo + Paclitaxel (N=75) | COHORT B Ipatasertib + Paclitaxel (N=145) | COHORT C Ipatasertib + Atezolizumab + Paclitaxel (N=102)
Anaemia (Blood and lymphatic system disorders) | 23 (34) | 43 (58) | 15 (28) | 45 (57) | 34 (50)
Leukopenia (Blood and lymphatic system disorders) | 4 (11) | 7 (23) | 7 (16) | 8 (18) | 11 (49)
Neutropenia (Blood and lymphatic system disorders) | 20 (39) | 28 (92) | 18 (58) | 36 (95) | 25 (114)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 9 (11) | 2 (2) | 4 (4) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 15 (16) | 7 (9) | 11 (17) | 12 (13)
Abdominal pain upper (Gastrointestinal disorders) | 8 (10) | 16 (16) | 5 (7) | 15 (21) | 6 (6)
Constipation (Gastrointestinal disorders) | 31 (40) | 49 (56) | 26 (33) | 42 (54) | 13 (20)
Diarrhoea (Gastrointestinal disorders) | 28 (56) | 138 (477) | 29 (64) | 125 (461) | 86 (324)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 14 (18) | 4 (6) | 9 (11) | 6 (7)
Flatulence (Gastrointestinal disorders) | 1 (1) | 5 (6) | 4 (6) | 7 (7) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (4) | 4 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 22 (29) | 66 (106) | 17 (28) | 60 (94) | 42 (65)
Stomatitis (Gastrointestinal disorders) | 6 (12) | 18 (31) | 6 (8) | 16 (27) | 7 (8)
Vomiting (Gastrointestinal disorders) | 8 (10) | 53 (112) | 6 (10) | 45 (67) | 28 (43)
Asthenia (General disorders) | 10 (12) | 35 (40) | 13 (17) | 27 (36) | 19 (22)
Fatigue (General disorders) | 15 (16) | 30 (33) | 19 (30) | 29 (36) | 23 (35)
Mucosal inflammation (General disorders) | 2 (4) | 11 (13) | 3 (4) | 8 (11) | 12 (12)
Oedema (General disorders) | 2 (2) | 5 (5) | 4 (4) | 9 (10) | 3 (3)
Oedema peripheral (General disorders) | 7 (7) | 18 (23) | 14 (19) | 21 (28) | 7 (9)
Pyrexia (General disorders) | 6 (6) | 16 (17) | 4 (5) | 23 (30) | 9 (13)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (12) | 0 (0) | 4 (38) | 6 (12) | 6 (13)
Hypersensitivity (Immune system disorders) | 5 (5) | 4 (8) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 3 (5) | 8 (9) | 6 (9) | 7 (12) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 11 (16) | 7 (11) | 19 (24) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 12 (13) | 6 (7) | 14 (19) | 8 (10)
Urinary tract infection (Infections and infestations) | 2 (3) | 12 (16) | 4 (7) | 16 (18) | 7 (9)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (8) | 6 (6) | 1 (1) | 6 (6) | 6 (12)
Alanine aminotransferase increased (Investigations) | 7 (16) | 23 (29) | 15 (30) | 19 (27) | 25 (59)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 18 (23) | 10 (16) | 13 (18) | 21 (39)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 9 (12) | 7 (9) | 3 (4) | 12 (20)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 7 (9) | 8 (11) | 5 (7) | 7 (10)
Neutrophil count decreased (Investigations) | 10 (23) | 22 (49) | 18 (65) | 23 (94) | 8 (33)
Weight decreased (Investigations) | 3 (3) | 12 (13) | 2 (2) | 7 (8) | 7 (7)
Weight increased (Investigations) | 1 (4) | 3 (4) | 3 (3) | 0 (0) | 6 (6)
White blood cell count decreased (Investigations) | 7 (15) | 11 (28) | 5 (27) | 10 (44) | 5 (10)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 29 (35) | 7 (15) | 21 (29) | 14 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (16) | 31 (49) | 10 (39) | 19 (27) | 22 (42)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (11) | 5 (8) | 7 (8) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (6) | 2 (2) | 6 (8) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (18) | 16 (24) | 10 (16) | 26 (40) | 13 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (14) | 16 (21) | 7 (8) | 21 (25) | 10 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (9) | 4 (4) | 9 (17) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 5 (6) | 3 (5) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 16 (24) | 9 (12) | 15 (17) | 10 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 14 (18) | 6 (6) | 13 (24) | 4 (5)
Dizziness (Nervous system disorders) | 8 (8) | 6 (8) | 3 (4) | 10 (12) | 10 (14)
Dysgeusia (Nervous system disorders) | 8 (8) | 10 (11) | 4 (4) | 11 (12) | 6 (6)
Headache (Nervous system disorders) | 10 (19) | 28 (56) | 8 (19) | 24 (37) | 21 (33)
Neuropathy peripheral (Nervous system disorders) | 20 (23) | 39 (49) | 12 (15) | 46 (63) | 30 (41)
Paraesthesia (Nervous system disorders) | 2 (3) | 8 (11) | 6 (8) | 13 (14) | 5 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 19 (19) | 32 (38) | 23 (24) | 23 (30) | 8 (8)
Polyneuropathy (Nervous system disorders) | 7 (7) | 5 (5) | 6 (6) | 12 (13) | 8 (8)
Insomnia (Psychiatric disorders) | 5 (6) | 10 (11) | 6 (6) | 6 (7) | 10 (10)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 9 (11) | 0 (0) | 3 (3) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 14 (15) | 6 (6) | 23 (32) | 16 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 7 (10) | 2 (2) | 10 (13) | 9 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 12 (14) | 4 (4) | 15 (17) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 13 (18) | 2 (3) | 11 (15) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 38 (39) | 78 (80) | 44 (46) | 75 (79) | 42 (42)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 5 (6) | 5 (5) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3) | 3 (4) | 5 (5) | 3 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (7) | 8 (8) | 9 (9) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 15 (21) | 3 (5) | 15 (25) | 17 (24)
Rash (Skin and subcutaneous tissue disorders) | 11 (13) | 26 (37) | 9 (13) | 31 (55) | 29 (40)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 4 (7) | 7 (7) | 5 (5)
Flushing (Vascular disorders) | 1 (2) | 3 (6) | 2 (2) | 4 (5) | 8 (8)
Hypertension (Vascular disorders) | 3 (3) | 6 (12) | 4 (7) | 8 (8) | 8 (9)
Lymphoedema (Vascular disorders) | 0 (0) | 7 (7) | 5 (6) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT03337724/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03337724/SAP_001.pdf